CLINICAL TRIAL: NCT02172573
Title: A Double-blind, Placebo-controlled, Randomised, Multicenter Trial to Compare the Safety and Efficacy of Oral Administration of Pramipexole up to 4.5mg and Bromocriptine up to 22.5mg Combined With L-dopa in Advanced Parkinson's Disease
Brief Title: Safety and Efficacy of Pramipexole and Bromocriptine Combined With L-dopa in Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 248.505
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Pramipexole; Bromocriptine

ARMS (3):
- Pramipexole (Experimental)
  Interventions: Drug: Pramipexole
- Bromocriptine (Experimental)
  Interventions: Drug: Bromocriptine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo pramipexole; Drug: Placebo bromocriptine

INTERVENTIONS:
Drug: Pramipexole
  Arms: Pramipexole
Drug: Bromocriptine
  Arms: Bromocriptine
Drug: Placebo pramipexole
  Arms: Placebo
Drug: Placebo bromocriptine
  Arms: Placebo

SUMMARY:
The objective of the study was to evaluate the efficacy and safety of SND 919 (pramipexole) tablets administered in combination with L-dopa in patients with Parkinson's disease using placebo and bromocriptine tablets as comparators in a double-blind design (phase III comparative study).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of Parkinson's disease (including juvenile parkinsonism)
* Patients who meet all of the following inclusion criteria

  * Patients who were at least 20 years of age
  * In- or outpatients of either sex
  * Patients in any stage on the modified Hoehn and Yahr scale
* Patients being treated with L-dopa who have any of the following clinical conditions and problems

  * Patients with the wearing-off phenomenon
  * Patients with the on-off phenomenon
  * Patients to whom a sufficient amount of L-dopa cannot be administered owing to the occurrence of an adverse event
  * Patients in whom the effect of L-dopa is attenuated
  * Patients in whom a dose increase of L-dopa has been refrained
  * Patients with freezing phenomenon

Exclusion Criteria:

* Patients being treated with other dopamine agonists (bromocriptine, pergolide mesylate, talipexole hydrochloride). Patients who have been treated with other dopamine agonist for at least 4 weeks before the start of the study (the day of giving informed consent) are eligible for the study
* Patients with a history of hypersensitivity to ergot preparations
* Patients with psychiatric symptoms such as confusion, hallucination, delusion, excitement, delirium, and abnormal behaviour
* Patients with subjective symptoms derived from orthostatic hypotension
* Patients with hypotension (systolic blood pressure less than 100 mmHg)
* Patients wiht Raynaud disease
* Patients with peptic ulcer
* Patients with complications such as severe cardiac, renal, hepatic disease etc.
* Patients with a current or past history of epilepsy
* Women who are or may be pregnant and lactating women
* Patients who are receiving any other investigational products or who have received any other investigational product within 6 months of the study
* Patients who are incompetent to give consent
* Others judged by the investigator or co-investigator to be ineligible as subjects

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 1999-04; Primary Completion 2000-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in total score of the Unified Parkinson's Disease Rating Scale (UPDRS) Part II (Activities of Daily Living) | Baseline and week 12
Change from baseline in total score of UPDRS Part III (Motor Examination) | Baseline and week 12

SECONDARY OUTCOMES:
Changes from baseline in sores of individual items on UPDRS Part II | Baseline and weeks 2, 4, 6, 8, 10, 12
Changes from baseline in scores of individual items on UPDRS Part III | Baseline and weeks 2, 4, 6, 8, 10, 12
Change from baseline in area under the curve (AUC) in the UPDRS Part II score | Baseline and weeks 2, 4, 6, 8, 10, 12
Change from baseline in area under the curve (AUC) in the UPDRS Part III score | Baseline and weeks 2, 4, 6, 8, 10, 12
Change from baseline in total score of UPDRS Part I (mentation, behaviour and mood) | Baseline and weeks 2, 4, 6, 8, 10, 12
Change from baseline in total score of UPDRS Part IV (complications of therapy) | Baseline and weeks 2, 4, 6, 8, 10, 12
Change from baseline in total score of UPDRS Part I-III | Baseline and weeks 2, 4, 6, 8, 10, 12
Change from baseline in total score of UPDRS Part I-IV | Baseline and weeks 2, 4, 6, 8, 10, 12
Change from baseline in Modified Hoehn & Yahr stage | Baseline and weeks 2, 4, 6, 8, 10, 12
Clinical global impression of efficacy | week 12
Number of patients with adverse events | up to 16 weeks
Number of patients with clinically significant changes in vital signs (blood pressure, pulse rate) | up to 12 weeks
Number of patients with abnormal changes in laboratory parameters | up to 12 weeks
Number of patients with abnormal changes in 12-lead electrocardiogram (ECG) | up to 12 weeks